CLINICAL TRIAL: NCT04522596
Title: Phase IV, Single-center, Double Blind, Randomized, Crossover, Placebo-controlled Study, to Investigate the Effect of Dual Bronchodilation With Umeclidinium Vilanterol on Patients With COPD, Hyperinflation and Heart Failure.
Brief Title: Effect of Dual Bronchodilation With Umeclidinium/Vilanterol on Patients With COPD, Hyperinflation and Heart Failure
Acronym: CHHEF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Luis Puente Maestu (Other)
Responsible Party: Sponsor-Investigator, Luis Puente Maestu, Professor, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHHEF; 2019-004427-20 (EudraCT Number)
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Copd; Heart Failure
Keywords: COPD; Heart failure; Hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — GSK573719; vilanterol

STUDY DESIGN:
Intervention Model Description: Phase IV clinical trial, single-center, double-blind, randomized, two-period crossover, placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Umeclidinium/vilanterol (Experimental): Umeclidinium/vilanterol 55/22 μg inhaled once a day for 14 days.
  Interventions: Drug: Umeclidinium/vilanterol
- Placebo (Placebo Comparator): Placebo inhaled once a day for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Umeclidinium/vilanterol — Umeclidinium/vilanterol 55/22 μg inhaled once a day
  Arms: Umeclidinium/vilanterol
Other: Placebo — Placebo inhaled once a day
  Arms: Placebo

SUMMARY:
Double-blind, randomized, two-period crossover, placebo-controlled, single-center study, to determine the effect of umeclidinium/vilanterol 55/22 μg compared with placebo on the increase in left systolic chamber function during exercise in patients with COPD, lung hyperinflation and mild to moderate left ventricular dysfunction.

DETAILED DESCRIPTION:
Phase IV clinical trial, single-center, double-blind, randomized, two-period crossover, placebo-controlled, to determine the effect of treatment with umeclidinium/vilanterol 55/22 μg compared with placebo on the increase in left systolic chamber function during exercise in patients with COPD, lung hyperinflation and mild to moderate left ventricular dysfunction.

The participants will be patients from the outpatient offices of the Cardiology, Pulmonology and Internal Medicine departments of the Gregorio Marañon University Hospital in Madrid, over 40 years of age with a diagnosis of COPD, lung hyperinflation with a residual volume more than 135 % and stable heart failure with a left ventricular ejection fraction between 35-55%.

Patients will be randomly assigned (1:1) to either umeclidinium/vilanterol 55/22 μg Ellipta for 14 days followed by a washout period of 14 days and then placebo for 14 days, or the same treatments in reverse order.

The randomization numbers will be generated by blocks of 4 elements selected with a computer-generated random list.

Patients, investigators, individuals in charge of the assessments, sponsor, CRO staff, and data analysts will be blinded to the identity and assignment of the treatments from the time of randomization until database lock, using the following methods:

1. Randomization data will be kept confidential until the time of unmasking (unlocking the database) and will not be accessible to anyone else involved in the study and
2. The identities of the treatments will be concealed by the use of active drugs and placebo identical in packaging, labeling, schedule of administration, appearance, and taste.

Two crossover treatment periods (treatments 1 and 2) of 14 days each separated by 14 days washout, and follow-up. The active treatment will be a combination of umeclidinium/vilanterol 55/22 μg Ellipta given by inhalation once per day over 14 days. Matching placebo will be used as a control. Any ongoing hypertensive and cardiovascular medications (including beta-blockers if prescribed) will be kept stable throughout the study. All previous COPD medications except inhaled corticosteroids (if dose stable for at least 30 days) will be withdrawn. Patients will be given salbutamol as rescue medication throughout the study and the respective study drugs in the treatment phases.

All adverse effects (AEs) spontaneously referred to either by the patients or during the visits will be registered and notified. All AEs will be collected, including those that are not considered associated with the study treatment.

All clinical information will be anonymously recorded in an e-CRF system programmed using in-house resources.

Any abnormal result of the study variables that the investigator considers clinically significant and require adjustments or transient or permanent interruption of treatment or any type of intervention or diagnostic evaluation to assess the associated risk for the patient will be collected as an adverse event and should be investigated and monitored adequately.

During the study, cardiac parameters will be determined by exercise echocardiography and MRI and assessed by experienced cardiologists (with cardiac MRI experience) blinded to all clinical and trial-related data.

Lung function will be assessed using constant-volume body plethysmography and spirometry in accordance with the American Thoracic Society and European Respiratory Society standards.

Patients will undergo a symptom-limited bicycle-exercise test at 30⁰ lateral decubitus in a dedicated ergometer (Easystress, Ecogito Medical SPRL, Liege, Belgium). Workrate will be initiated at 25 W and increased by 15 W every 3 min. The gas exchange will be simultaneously analyzed breath-by-breath (Ergostik, Geratherm, Germany). Doppler-derived stroke volume, systolic ejection period, and left ventricular outflow tract, at a specific point from the aortic valve, will be measured as recommended. The LV outflow tract cross-sectional area will be assumed constant so that the change in SV will be determined by the change in the outflow tract time-velocity integral as measured by pulsed-wave Doppler. We have recently validated the Doppler-derived method for measuring SV during exercise.

Baseline LV volumes and ejection fraction will be measured using the biplane Simpson's method. In addition, color-Doppler M-mode images will be acquired at baseline and during all exercise phases both for the ejection and diastolic phases at the outflow and inflow tract locations, respectively. These recordings have been validated both in clinical and preclinical studies as robust and load-independent indices of global LV systolic chamber function and diastolic suction, respectively. Furthermore, the ejection intraventricular pressure difference (EIVPD) is a simple but very sensitive method to detect subtle changes in LV systolic function, undetectable by other conventional methods.

Because frequently patients do not reach the anaerobic threshold during exercise echocardiography (decubitus…), a separate maximal ergospirometry on a cycle ergometer will be performed to measure peak exercise capacity. The cycle ergometer (ER-900, Vyasis, Hochberg, Germany) exercise test will start with a period of quiet breathing for at least 3 min followed by unloaded pedaling for 3 min, thereafter an immediate increase in work rate to 10 W and then by further increments of 10 W every minute until symptom limitation during which breath by breath gas exchange ( i.e. VO2 and VCO2) (Oxycon-pro Vyasis, Hoechberg Germany) lactate threshold (if attained by the patient) maximum ventilation and heart-rate dyspnea, inspiratory capacity and exercise flow-volume loops (every 2 min) and HR recovery rate will be measured. Peak oxygen uptake will be defined as the greatest work rate that was maintained for ≥30 s at 50-70 rpm.

Patients will undergo a conventional cardiac MRI study (Philips Achieva 1.5 T) without gadolinium to assess the size of the left and right ventricles. In addition, phase-contrast studies will be obtained to address cardiac output and flow characteristics at the level of the aorta and the main pulmonary artery, as previously described.

Patient reported outcomes will be assessed using the COPD assessment test (CAT) to measure health status and the transition dyspnea index to measure dyspnea.

External data monitorization and Adverse Event Reporting shall be contracted to an independent CRO, following current standards of clinical investigation

Primary objective:

To address the effect (compared with placebo) of umeclidinium/vilanterol 55/22 μg on the increase in exercise stroke volume (from baseline).

Secondary objectives:

To address the effect (compared with placebo) of umeclidinium/vilanterol 55/22 μg on the reduction of dynamic hyperinflation (from baseline).

To address the effect (compared with placebo) of umeclidinium/vilanterol 55/22 μg on resting cardiac function (from baseline).

To address the effect (compared with placebo) of umeclidinium/vilanterol 55/22 μg on PROMs (patient-reported outcomes measurement) from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 85 years with a clinical diagnosis of COPD
* Airflow limitation indicated by a screening post-bronchodilator FEV1 < 80% and >35% predicted and a post-bronchodilator FEV1/FVC < 0.7
* Smoking history of at least ten pack-years
* Baseline lung hyperinflation with a residual volume of more than 135% predicted
* Stable heart failure
* Left ventricle ejection fraction in the range of 35% to 55%.
* A suitable ultrasonic window from the apical view
* No exacerbation within 2 months before study recruitment (defined as the use of systemic corticoids, antibiotics, or hospitalization)

Exclusion Criteria:

* Do not sign the informed consent
* Unstable cardiovascular diseases
* Atrial fibrillation or other arrhythmias requiring treatment
* Unstable ischemic heart disease
* Uncontrolled hypertension
* Patients unable to undergo cardiac MR scanning (claustrophobia or carrying non-MR-compatible devices)
* Patients unable to perform an exercise test (locomotor conditions)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the increase in exercise stroke volume. | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Baseline-corrected, time-velocity integral (a direct surrogate of SV) during peak exercise, as measured by exercise Doppler-echocardiography.
Change from baseline on the increase in exercise oxygen pulse. | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Maximal oxygen pulse on a cardiopulmonary exercise test on Cycle-ergometer

SECONDARY OUTCOMES:
Change from baseline on the reduction of resting hyperinflation.. | Screening (-14), 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Resting lung volumes (Inspiratory capacity, functional residual capacity and residual volume)
Change from baseline on the reduction of dynamic hyperinflation. | Screening (-14), 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Inspiratory Capacity every 2 minutes during the incremental exercise test.
Change from baseline on resting dyastolic left heart function. | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Left and right cardiac chambers volumes at rest in patients, as measured by MRI (Baseline)
Change from baseline on resting systolic left cardiac function. | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Baseline-corrected peak ejection intraventricular pressure difference (peak EIVPD) at peak exercise, as measured by exercise color-Doppler M-mode echocardiography.
Change from baseline on resting right cardiac function. | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Pulmonary acceleration time in the main pulmonary artery as measured by phase-contrast MRI.
Change from baseline on resting left cardiac function. | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Baseline-corrected peak intraventricular diastolic pressure gradient (peak DIVPD) at peak exercise - diastolic suction, as measured by exercise color-Doppler M-mode echocardiography.
Change from baseline on PROMs (Impact of disease). | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Average changes in COPD Assessment Test (CAT)
Change from baseline on PROMs (dyspnea). | 0, 14, 42 days (Visits 4, 5 and 7 respectively)
  Proportion of patients with Clinically relevant changes in Transition dyspnea index ( -4 and -2 respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Puente-Maestu, Prof, Study Director — Instituto de Investigación Sanitaria Gregorio Mrañón
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain